CLINICAL TRIAL: NCT02410226
Title: Comparison Between Ultrasound-assisted and Conventional Palpation Techniques for Epidural Catheterization Before Cesarean Section
Brief Title: Ultrasound Versus Palpation for Epidural Catheterization
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Mohamed Mohamed Tawfik, Lecturer, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: R115
Record Dates: First submitted 2015-03-30; First posted 2015-04-07 (Estimated); Last update posted 2015-09-23 (Estimated); Status verified 2015-09

CONDITIONS: Epidural Anesthesia; Spinal Ultrasound

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Palpation (Active Comparator): Double-space combined spinal-epidural anesthesia, Sham ultrasound procedure
  Interventions: Procedure: Double-space combined spinal-epidural anesthesia; Radiation: Sham ultrasound procedure
- Ultrasound (Experimental): Double-space combined spinal-epidural anesthesia, Preprocedure spinal ultrasound
  Interventions: Procedure: Double-space combined spinal-epidural anesthesia; Radiation: Preprocedure spinal ultrasound

INTERVENTIONS:
Procedure: Double-space combined spinal-epidural anesthesia — Epidural space identification in Lumbar 2-3 or 3-4 space using loss of resistance to air technique with 18-gauge Tuohy needle, then threading a 20-gauge multi-orifice epidural catheter 4-5 cm into the epidural space. Spinal anesthesia administration in an appropriate lower intervertebral space with intrathecal bupivacaine 12.5 mg and fentanyl 10 mcg through a 27-gauge spinal needle.
Radiation: Preprocedure spinal ultrasound — Lumbar spinal ultrasound using the 2-5 MHz curved probe, performed in both the longitudinal and transverse planes for identification of the appropriate intervertebral spce, estimation of the depth to the epidural space, and noting the proper angle for subsequent needle insertion. Then skin markings relying on the ultrasound procedure are made identifying 2 intervertebral spaces.
  Arms: Ultrasound
Radiation: Sham ultrasound procedure — Applying the ultrasound probe on the patient's back while the ultrasound machine is on the freeze position.Then skin markings relying on landmark palpation are made identifying 2 intervertebral spaces.
  Arms: Palpation

SUMMARY:
The study will assess the benefit of using spinal ultrasound before epidural catheter insertion compared to the conventional palpation technique in women undergoing cesarean section.

DETAILED DESCRIPTION:
The study will compare the ultrasound-assisted and the conventional palpation techniques for epidural catheterization as a component of combined spinal-epidural anesthesia for cesarean section.

Participants will be randomly assigned into 2 equal groups. In the ultrasound group: Preprocedure lumbar spinal ultrasound will be performed before epidural catheterization. In the palpation group: Conventional technique of landmark palpation will be used.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists class I or II.
* Full term parturients scheduled for elective cesarean delivery under combined spinal-epidural anesthesia.

Exclusion Criteria:

* Body mass index ≥ 35 kg/m2.
* Patients having any contraindication to neuraxial anesthesia (Refusal of the procedure, Coagulopathy, Uncorrected hypovolemia, Increased intracranial pressure, Local skin infection).
* Marked spinal deformity or previous spinal surgery.
* Unpalpable anatomical landmarks.
* Emergent situations.

Ages: 19 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 110 (Actual)
Dates: Start 2015-04; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Rate of successful epidural catheterization at the first needle pass | 24 hours after delivery
  Needle pass includes any forward advancement of the Tuohy needle.

SECONDARY OUTCOMES:
Rate of successful epidural catheterization at the first skin puncture | 24 hours after delivery
  Skin puncture includes any separate skin puncture by the Tuohy needle.
Number of needle passes required for successful epidural catheterization | 24 hours after delivery
Number of skin punctures required for successful epidural catheterization | 24 hours after delivery
Time of the epidural catheterization procedure | 24 hours after delivery
  From the initial Tuohy needle insertion through the skin to the completion of the threading of the epidural catheter.
Patient satisfaction (5-point scale) | 24 hours after delivery
  5-point scale
Rate of Inadvertent dural puncture | 24 hours after delivery
Rate of Inadvertent vascular puncture | 24 hours after delivery
Rate of Failed block | At the first request of analgesia
  Complete failure of epidural catheter after 2 doses of epidural injection of 10 ml bupivacaine 0.25% and fentanyl 20 mcg administered 20 min apart.
Unilateral / Patchy block (Assessed by pinprick) | At the first request of analgesia
  Assessed by pinprick after 20 min of epidural injection of 10 ml bupivacaine 0.25% and fentanyl 20 mcg
Rate of Back pain | 24 hours after delivery

OTHER OUTCOMES:
Level of successful epidural catheterization | 24 hours after delivery
  The lumbar intervertebral space L 2-3 or 3-4 used for epidural catheter insertion.

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed M Tawfik, M.Sc., Principal Investigator — Department of Anesthesia and Surgical Intensive Care, Mansoura University Hospitals.
Locations (1):
- Department of Anesthesia, Mansoura University Hospitals, Al Mansurah, Dakahlia Governorate, Egypt